CLINICAL TRIAL: NCT06829433
Title: Quantifying the Movement Dynamics of Adults Living With Total Knee Arthroplasty and Knee Osteoarthritis
Brief Title: Movement Dynamics of Knee Osteoarthritis and Total Knee Replacement
Acronym: MDOA&TKR
Status: Recruiting | Type: Observational
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Josie Morris, Principal Investigator, University of Portsmouth
Other Study IDs: SHFEC 2024-007
Record Dates: First submitted 2025-01-28; First posted 2025-02-17 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Total Knee Replacement
  Interventions: Other: No intervention
- Knee Osteoarthritis
  Interventions: Other: No intervention
- Asymptomatic Controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational cross-sectional study

SUMMARY:
This research aims to explore differences in walking and functional movement mechanics, exercise response, and physical activity between people with osteoarthritis (OA), those who have undergone total joint replacement, and healthy individuals.

DETAILED DESCRIPTION:
People living with OA tend to be less physically active than those without the disease, which is often due to pain, stiffness and joint instability. This reduction in physical activity can lead to additional health problems down the line. When the disease becomes severe, joint replacement surgeries are sometimes performed to relieve pain and improve individuals' quality of life. However, despite reducing pain, there is little evidence to show that joint replacement surgeries encourage individuals to return to healthy physical activity levels.

Reasons for the lack of change may include a failure to address unhealthy walking and movement patterns which could still be causing pain and instability and reduced physical fitness levels.

By investigating these reasons, we hope that findings from this study will help to inform future interventions that improve clinical outcomes and quality of life for individuals with OA and post-joint replacement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed symptomatic bilateral or unilateral knee osteoarthritis, self-reported ability to walk without an aid for 10 minutes and to ascend and descend stairs, no neurological conditions or other musculoskeletal pathology/injury which would impact walking gait.

Exclusion Criteria:

* Unable to walk at 0.8 m/s, exclusion based on IMO screening, non-English speaking, lacking ability to consent.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Local private physiotherapy clinics and local sports clubs
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Peak knee adduction moment | From the start of a biomechanical movement testing visit to the end (approximately 2 hours)
  The external knee adduction moment (KAM), which reflects medial-to-lateral knee joint load distribution during gait, has become an OA treatment target. The peak KAM is a strong predictor of presence, severity, and the rate of progression of knee OA.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychology, Health and Sport Sciences, University of Portsmouth, Portsmouth, Hampshire, United Kingdom